CLINICAL TRIAL: NCT03290963
Title: Targeting mTOR/GSK3 With Lithium Augmentation to Enhance and Sustain Rapid Antidepressant Actions of Ketamine in Adults With Treatment-Resistant Depression: A Precision Medicine Approach for Psychiatry
Brief Title: Effect of Lithium Versus Placebo in Adults With Treatment-Resistant Depression Who Are Receiving Ketamine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator moved to Jacksonville, FL campus.
Sponsor: William V. Bobo, M.D. (Other)
Responsible Party: Sponsor-Investigator, William V. Bobo, M.D., Professor of Psychiatry, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 17-000819
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Treatment Resistant Depression
Keywords: depression; bipolar I disorder; bipolar II disorder
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression; Bipolar Disorder | interventions — Lithium; Lithium Carbonate; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple blinded study. The staff accessible to the blind includes pharmacy staff and one assigned investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine plus Lithium (Active Comparator): Lithium will be used in conjunction to Ketamine infusions for the treatment of major depression disorder or bipolar disorder type I or II. Before the first ketamine infusion, subjects will be randomized to 2 weeks of lithium treatment. All subjects will receive three IV ketamine infusions (0.5 mg/kg, over 100 min.) over 7 days. Those who achieve positive response (>50% decrease in MADRS total score from baseline) will be given 4 additional once-weekly ketamine infusions (same dose and infusion rate) and lithium treatment .
  Interventions: Drug: Lithium; Drug: Ketamine
- Ketamine plus Placebo (Placebo Comparator): Placebo tablets will be used in conjunction to Ketamine infusions for the treatment of major depression disorder or bipolar disorder type I or II. Before the first ketamine infusion, subjects will be randomized to 2 weeks of placebo treatment. All subjects will receive three IV ketamine infusions (0.5 mg/kg, over 100 min.) over 7 days. Those who achieve positive response (>50% decrease in MADRS total score from baseline) will be given 4 additional once-weekly ketamine infusions (same dose and infusion rate) and placebo treatment.
  Interventions: Drug: Placebo; Drug: Ketamine

INTERVENTIONS:
Drug: Lithium — Lithium will be dosed in units (LI level > or = 0.4 milliequivalents (mEq)/L)
  Other Names: Lithane; Lithobid
  Arms: Ketamine plus Lithium
Drug: Placebo — Placebo tablets, dosed in units
  Arms: Ketamine plus Placebo
Drug: Ketamine — All subjects will receive 3 IV ketamine infusions of 0.5mg/kg, over 100 min. over 7 days.
  Other Names: Ketalar

SUMMARY:
The purpose of this research study is to compare the antidepressant effect of lithium versus placebo in adults receiving ketamine. Lithium is available commercially for depression; ketamine is available commercially and can help the symptoms of depression; however, it has not been approved by the U.S. Food and Drug Administration (FDA) for this use. The FDA has allowed the use of this drug in this research study.

DETAILED DESCRIPTION:
This is a randomized clinical trial in adults with Treatment-Resistant Depression. All participants will receive three intravenous (IV) Ketamine (KET) infusions over 7 days. Before receiving the first KET infusion, subjects will be randomized to 2 weeks of pre-KET treatment with either Lithium or matching placebo. Pre-treatment medications will then be continued in a double-blind manner during the acute phase administration of ketamine. Questionnaires will be administered at baseline, prior to each KET infusion, and at 40, 100, and 120 minutes after each infusion, and again at weekly intervals following the third (final) KET infusion for 4 weeks, using standardized rating scales. Those who achieve positive response (>50% decrease in questionnaire total score from baseline) will be given 4 additional once-weekly KET infusions (same dose and infusion rate).

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent;
* Current psychiatric inpatient (voluntary only) or outpatient treatment;
* Meets Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) diagnostic criteria for major depressive disorder, bipolar I disorder, or bipolar II disorder;
* 9-item Patient Health Questionnaire (PHQ-9) total score > 15 at screening and at baseline (just prior to first acute phase ketamine infusion);
* Treatment-resistant depression, as defined by failure of at least two previous antidepressant or mood stabilizing treatments within the current depressive episode. Failed antidepressant or mood stabilizing treatments can include pharmacotherapy for depression at an adequate dose for at least 8 weeks, or an acute series of at least 6 administrations of electroconvulsive therapy (ECT);
* Adequate social support, defined as having at least one individual identified who is committed to function as support, including providing transportation to and from outpatient ketamine infusion visits;
* Ability to pass a comprehension assessment test related to effects of ketamine and trial objectives and criteria.

Exclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder, or active psychotic symptoms;
* On active lithium treatment;
* Serious risk for suicide, as assessed by the evaluating study clinician; a serious suicide risk will be considered: (a) an inability to control suicide impulses or imminent or unacceptably high risk of suicide in the investigator's judgment; or (b) a recent history of suicidal behavior, which is defined as either one or more suicide attempts (or interrupted suicide attempts) in the 12 months before study entry; or (c) history of serious suicidal behavior, defined as one or more suicide attempts (or interrupted attempts) in the last 3 years with a potential lethality judged by the evaluating study clinician to have possibly resulted in serious injury or death;
* Ongoing prescription of > 4 mg lorazepam equivalents (total) daily, or morning dosing of any benzodiazepine at the time of assessment;
* Currently undergoing ECT, transcranial magnetic stimulation, vagal nerve stimulation, or deep brain stimulation as either an acute or maintenance treatment of depression;
* Any active or unstable medical condition judged by the study psychiatrist as conferring too great a level of medical risk to allow inclusion in the study;
* Use or abuse of methamphetamine, cocaine, cannabis, or stimulants (prescribed and illicit) within the past 12 months;
* Any current abuse or dependence of alcohol or drugs (excluding nicotine and caffeine). Note: Persons will be allowed to enroll in this study if their drug or alcohol abuse/dependence is in complete (not partial) and sustained (> 1 year) remission;
* History of traumatic brain injury that resulted in loss of consciousness;
* Developmental delay, mental retardation, or intellectual disorder;
* Clinical or self-reported diagnosis of delirium, encephalopathy, or related clinical diagnosis within the prior 12 months;
* Cognitive disorder (mild and major categories, per DSM-5);
* Prior participation in another study of ketamine for depression within the prior 6 months;
* History of either poor antidepressive response to or poor tolerability of ketamine (any route of administration) when previously administered for treating symptoms of depression;
* History of hypothyroidism unless taking a stable dose of thyroid medication and asymptomatic for 6 months;
* Significant unstable medical condition
* Hepatic insufficiency (2.5 X Upper Limit of Normal (ULN) for Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT)) within 1 year of consent, past liver transplant recipient, and/or clinical diagnosis of cirrhosis of the liver;
* History of either poor antidepressive response to or poor tolerability of ketamine (any route of administration) when previously administered for treating symptoms of depression;
* History of medical condition(s) which are not recommended to be taken concurrently with lithium; Current anti-depressive pharmacotherapies will not be allowed during the acute phase KET infusions.
* Pregnancy, or nursing;
* Prisoners;
* Involuntary psychiatric hospitalization.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | baseline, at the end of the first infusion (approximately 1 day)
  The Montgomery Asberg Depression Scale (MADRS) is a 10-item observer rating scale assessing symptoms of depression. The score ranges from 0 (no depression) to 60 (very depressed).
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | baseline, at the end of third infusion (approximately 7 days)
  The Montgomery Asberg Depression Scale (MADRS) is a 10-item observer rating scale assessing symptoms of depression. The score ranges from 0 (no depression) to 60 (very depressed).

CONTACTS AND LOCATIONS:
Overall Officials: William V Bobo, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No